CLINICAL TRIAL: NCT02386943
Title: An Open-label, Randomized,Three-way Cross-over, Single Dose Study to Explore the Effect of DPP-4 Inhibitors on β-cell Function by Using the Two-step Hyperglycemic Clamp
Brief Title: Study on Exploring the Effect of DPP-4 Inhibitors on β-cell Function by Using the Two-step Hyperglycemic Clamp
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Shanghai Jiao Tong University Affiliated Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD022
Record Dates: First submitted 2015-03-07; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; saxagliptin; BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin (Experimental): Subjects are assigned to take one pill of sitagliptin(100mg po once) at 7am on experimental day,then the two-step hyperglycaemic clamp is initiated at 9am.
  Interventions: Drug: Sitagliptin
- Saxagliptin (Experimental): Subjects are assigned to take one pill of saxagliptin(5mg po once) at 7am on experimental day,then the two-step hyperglycaemic clamp is initiated at 9am.
  Interventions: Drug: Saxagliptin
- Blank control (Experimental): Subjects take no medication for blank control at experimental day,then the two-step hyperglycaemic clamp is initiated at 9am.
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Sitagliptin — 100mg po once.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Saxagliptin — 5mg po once.
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Blank control — No medication is taken.
  Other Names: Baseline
  Arms: Blank control

SUMMARY:
The objective of this study is to explore the effects of two DPP-4 inhibitors(Sitagliptin, Saxagliptin) on β- and α-cell function, as well as the incretin effect.

DETAILED DESCRIPTION:
The study is an open-label, randomized, three-way crossover and single-dose study.Subjects with newly onset T2DM are enrolled. They are assigned to take a single dose of sitagliptin (100 mg), saxagliptin (5 mg), or blank control in a randomized order separated by a washout period of 7-14 days.Then the two-step hyperglycemic clamp is initiated.

On each experimental day, the subject will take the given dose of Sitagliptin, Saxagliptin and nothing for blank control two hours before the clamp experiment starts.

The hyperglycaemic clamp will be performed after an overnight fast. Subjects will be placed in a recumbent position and cannula will be inserted in a dorsal hand vein. The hand will be placed in a heating box (50℃) throughout the experiment to allow frequent sampling of arterialized blood. A second cannula will be inserted in a contralateral cubital vein for glucose infusion.

At time zero (0 min), a 50% glucose bolus will be injected during 1 min to increase PG to 15mM. The glucose bolus will be calculated as:(15mM-FPG)×35 mg glucose × body weight (kg). PG will be measured bedside every 5 min and maintained at 15mM by an adjustable continuous 20% glucose infusion. After 90min, PG will be lowered down to 7mM for the islet cells to rest, then the subject will be instructed to consume 75g glucose solution orally in 5min. 40min after the oral glucose consumption, the 90min-hyperglycaemic clamp experiment wil be restarted. The oral period of hyperglycaemic clamp process is the same as what's done in fasting period. Blood samples will be collected in -2h, 0min, 10min, 90min in both hyperglycaemic clamp experimental process for the measurement of insulin, c-peptide, glucagon, active GLP-1 and other incretin hormones.

Thus we could evaluate the beta cell function represented by the first phase and the second phase of insulin secretion(C-peptide secretion) and alpha cell function represented by the change of glucagon concentration during the fasting period and oral period of hyperglycaemic clamp experiment and the change of active GLP-1.

ELIGIBILITY:
Inclusion Criteria:

1. 40-60 years old;
2. Diagnosed as T2DM according to the 1999 World Health Organization criteria within 2 years;
3. Free of any antihypoglycemia therapy ever;
4. No weight fluctuation greater than 5% in late 3 months.
5. Understand and voluntarily sign an informed consent document.
6. Good study compliance.

Exclusion Criteria:

1. With any significant medical condition (within 3 years), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study;
2. Used any prescribed systemic or topical medication within 30 days of the first dose administration;
3. Any medical or surgical conditions possibly affecting study drug absorption, distribution, metabolism and excretion;
4. Participated in a clinical study involving administration of an investigational drug within 90 days preceding the first dose administration or within five half-lives of the first dose administration (whichever is longer);
5. Donated blood or plasma or had any other significant blood loss within 2 months preceding the first dose administration;
6. History of multiple drug allergies;
7. Any clinically significant allergic disease;
8. Recently drug or alcohol abuse (>35 unit/week, 1 unit=8g alcohol @ 1 standard drink @ 250ml beer @ 140ml wine @ 25ml strong alcohol drink like whiskey); Smokers or users of other tobacco products in the 3 months prior to screening.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
β-cell function (measurement of insulin and c-peptide during the clamp study) | 15 months
  The primary endpoints are the effects of DPP-4 inhibitors on β-cell function, with the measurement of insulin and c-peptide during the clamp study.

SECONDARY OUTCOMES:
α-cell function (measurement of glucagon during the clamp study) | 15 months
  The secondary endpoints are the effects of DPP-4 inhibitors on α-cell function, with the measurement of glucagon during the clamp study.
Incretin effect (measurement of active GLP-1 during the clamp study) | 15 months
  The secondary endpoints are the effects of DPP-4 inhibitors on incretin effect, with the measurement of active GLP-1 during the clamp study.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, China